CLINICAL TRIAL: NCT01411813
Title: Alprazolam and Eating Behavior in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #6267; 5R01MH082736 (NIH)
Record Dates: First submitted 2011-04-15; First posted 2011-08-08 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alprazolam: Patients receiving Alprazolam.

SUMMARY:
This study examines the role of anxiety in food intake among patients with AN by measuring caloric intake in a standardized, laboratory meal with alprazolam versus a placebo. Patients will participate in two test meal sessions, one after receiving alprazolam and one after receiving a placebo. Patients will be administered psychological measures of anxiety, mood, and eating behavior. Primary outcomes include caloric intake in a laboratory test meal and pre-meal anxiety levels.

DETAILED DESCRIPTION:
30 patients with Anorexia Nervosa (hospitalized at NYSPI 4-Center for acute weight restoration treatment) will be recruited to participate in this experiment. All subjects will be screened on admission and provide informed consent prior to participation. At the time of study procedures, participants will be medically stable and weigh ≥ 80% IBW. This minimum weight has been identified for patient safety given the test meal procedures. Subjects will participate in a total of two meal sessions on the BSU. Medical clearance will be determined by 4-Center clinical staff prior to the meal sessions. Study participation will not prolong nor interfere with the patient's treatment.

The first test meal will occur after the patient has reached 80% IBW. The second test meal will occur within a week of the first. The procedures are identical for the two test sessions, and were based on those described by Sysko and colleagues (9). On the morning of the test meal, participants will be provided a standardized breakfast of ~300 kcal. They will not consume any additional food or liquid, other than water, prior to the test meal session approximately 4 hours later. Study medication will be administered at 10:00 am.

Test meals will be conducted on the Biological Studies Unit (BSU) at NYSPI. Participants will be escorted to and from the BSU by research staff. Participants will complete questionnaires prior to receiving medication, prior to each test meal, and after the test meal is complete (see Table). Participants will be presented with an 83 fluid ounce covered opaque container with a straw on a table. Inside the container will be approximately 1500 grams (approximately 1560 kcal) of strawberry yogurt shake. Patients will be informed that the meal consists of a strawberry yogurt shake, but will not be informed as to the amount provided in the container. Instructions before each test meal will inform patients that they should eat as much of the shake as they would like, and that the meal would serve as their lunch for the day. The participant will be alone in the room. For compliance and safety, patients will be observed through a closed circuit video monitor during the meal. The patient will be instructed to signal completion of the meal by ringing a bell. During the course of the meal, patients will be asked to rate anxiety periodically. After the test meal is complete, a staff member will debrief the participant and address any questions or concerns.

Medication Administration: Participants will receive active medication (alprazolam 0.75 mg) on one test day and placebo on the other, in random order. Dose was selected based on the findings of Evans et al (8), who demonstrated statistically significant increases in caloric intake with doses of alprazolam 0.5 mg and 0.75 mg. Medication will be administered 2 hours prior to the test meal, as this is the timing of estimated peak plasma concentration (8).

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR™ diagnosis of anorexia nervosa (restricting or binge-purge subtype), with or without amenorrhea at the time of inpatient admission.
2. Older than 18
3. No acute medical condition
4. Participation in inpatient treatment
5. Subjects must have signed informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Psychotic or bipolar I disorder
2. Substance abuse or dependence in the last 6 months
3. Current Axis I disorder requiring psychotropic medication (subjects taking a stable dose of psychiatric medications will be allowed.)
4. Active suicidal intent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Anorexia Nervosa hospitalized at NYSPI 4-C unit
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change in caloric Intake | Change in caloric intake between test meals
  Assessment of caloric intake after taking alprazolam or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Steinglass, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Steinglass JE, Kaplan SC, Liu Y, Wang Y, Walsh BT. The (lack of) effect of alprazolam on eating behavior in anorexia nervosa: a preliminary report. Int J Eat Disord. 2014 Dec;47(8):901-4. doi: 10.1002/eat.22343. Epub 2014 Aug 19. PMID 25139178